CLINICAL TRIAL: NCT00785863
Title: Modulation of Remifentanil-induced Analgesia and Postinfusion Hyperalgesia by Parecoxib or Ketorolac in Humans
Brief Title: Modulation of Remifentanil-induced Postinfusion Hyperalgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other); Rikshospitalet University Hospital (Other)
Responsible Party: Ullevaal University Hospital, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2008-000904-10
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2008-11

CONDITIONS: Hyperalgesia, Secondary
Keywords: hyperalgesia; remifentanil; ketorolac; parecoxib; COX-1 inhibitor; COX-2 inhibitor
MeSH Terms: conditions — Hyperalgesia | interventions — Remifentanil; Ketorolac; Ketorolac Tromethamine; parecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Remifentanil (Active Comparator)
  Interventions: Drug: Remifentanil
- Ketorolac and remifentanil (Active Comparator)
  Interventions: Drug: Ketorolac and remifentanil
- Parecoxib and remifentanil (Active Comparator)
  Interventions: Drug: Parecoxib and remifentanil

INTERVENTIONS:
Other: Placebo — Placebo IV before placebo infusion
  Arms: Placebo
Drug: Remifentanil — placebo IV and remifentanil infusion
  Other Names: Ultiva
  Arms: Remifentanil
Drug: Ketorolac and remifentanil — Ketorolac IV and remifentanil infusion
  Other Names: Toradol
  Arms: Ketorolac and remifentanil
Drug: Parecoxib and remifentanil — Parecoxib IV and remifentanil infusion
  Other Names: Dynastat
  Arms: Parecoxib and remifentanil

SUMMARY:
In addition to alleviate pain there is growing evidence that µ-opioids enhance pain. This problem is known as opioid induced hyperalgesia(OIH).The NMDA receptor is involved in opioid induced hyperalgesia it may be possible to block OIH by cyclooxygenase inhibitors. This has been demonstrated with parecoxib, a COX-II inhibitor, in a experimental pain model.Both COX-1 and COX-2 are expressed in the spinal cord. It would be of interest to investigate whether a COX-1 preferring inhibitor like ketorolac also can reduce opioid induced hyperalgesic in this experimental pain model.

DETAILED DESCRIPTION:
Remifentanil is an fast acting opioid which has become very popular to use during surgery.

There are studies, both experimental 1-3 and clinical 4;5, which indicate that remifentanil after end of infusion trigger enhanced pain experience and enhanced opioid consumption postoperatively.

Therefore it is important to look at possibilities to block this enhanced pain experience (opioid induced hyperalgesia - OIH). Ketamin has demonstrated to block this effect 5;6 through the NMDA receptor. Unfortunately ketamin has some seriously side-effects like hallucinations, and is therefore not suitable in ordenary clinical use.

Recently, it has been demonstrated that parecoxib (a COX-2 inhibitor) can prevent remifentanil-induced postinfusion hyperalgesia in a study on healthy volunteers.7 COX-2 inhibitors have some disadvantages because of the longterm adverse effects like cardiac arrest. Therefore it would be of interest to look at a COX-1 preferring NSAID, like ketorolac, to see if also non-selective NSAIDs can partly block remifentanil-induced postinfusion hyperalgesia.

To investigate this and to provoke pain and secondary hyperalgesia we use an intradermal electrical pain model which is well established.1;7-9 Detailed description of this model look at reference 7. H0 : Parecoxib prevents remifentanil postinfusion secondary hyperalgesi. Ketorolac does not prevent remifentanil postinfusion secondary hyperalgesi HA : Parecoxib and ketorolac prevent remifentanil postinfusion secondary hyperalgesi.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Allergy to the drugs used in the study

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
H0 : Parecoxib prevents remifentanil postinfusion secondary hyperalgesi. Ketorolac does not prevent remifentanil postinfusion secondary hyperalgesi. | during the study

SECONDARY OUTCOMES:
HA : Parecoxib and ketorolac prevent remifentanil postinfusion secondary hyperalgesi. | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Harald Lenz, MD, Principal Investigator — Ullevaal University Hospital; Johan Raeder, Prof.,MD,PhD, Study Director — Ullevaal University Hospital; Audun Stubhaug, Prof.,MD,PhD, Study Director — Rikshospitalet University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Oslo County, Norway